CLINICAL TRIAL: NCT00507416
Title: Randomized Phase 3b Study of Three Treatment Regimens in Subjects With Previously Untreated Multiple Myeloma Who Are Not Considered Candidates for High-Dose Chemotherapy and Autologous Stem Cell Transplantation: VELCADE, Thalidomide, and Dexamethasone Versus VELCADE and Dexamethasone Versus VELCADE, Melphalan, and Prednisone
Brief Title: Velcade,Thalidomide, and Dexamethasone Versus Velcade and Dexamethasone Versus Velcade, Melphalan, and Prednisone
Acronym: UPFRONT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C05009
Record Dates: First submitted 2007-07-25; First posted 2007-07-26 (Estimated); Results first posted 2014-05-01 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2014-03

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Dexamethasone; Melphalan; Prednisone; Thalidomide

ARMS (3):
- Bortezomib and Dexamethasone (VD) (Experimental): Participants received bortezomib (Velcade) 1.3 mg/m^2 administered as a bolus intravenous (IV) injection on Days 1, 4, 8, and 11, and dexamethasone 20 mg orally on Days 1, 2, 4, 5, 8, 9, 11 and 12 for eight 21-day treatment cycles (Induction). Participants then received bortezomib 1.6 mg/^2 IV on Days 1, 8, 15 and 22 for five 35-day cycles (Maintenance).
  Interventions: Drug: Bortezomib; Drug: Dexamethasone
- Bortezomib, Thalidomide, and Dexamethasone (VTD) (Experimental): Participants received bortezomib (Velcade) 1.3 mg/m^2 administered as a bolus IV injection on Days 1, 4, 8, and 11, and dexamethasone 20 mg orally on Days 1, 2, 4, 5, 8, 9, 11 and 12, and thalidomide 100 mg orally on Days 1-21 for eight 21-day treatment cycles (Induction). Participants then received bortezomib 1.6 mg/^2 IV on Days 1, 8, 15 and 22 for five 35-day cycles (Maintenance) .
  Interventions: Drug: Bortezomib; Drug: Dexamethasone; Drug: Thalidomide
- Bortezomib, Melphalan and Prednisone (VMP) (Experimental): Participants received bortezomib (Velcade) 1.3 mg/m^2 administered as a bolus IV injection on Days 1, 4, 8, and 11, and melphalan 9 mg/m^2 orally on Days 1-4 every other cycle and prednisone 60 mg/m^2 orally on Days 1-4 every other cycle for eight 21-day treatment cycles (Induction). Participants then received bortezomib 1.6 mg/^2 IV on Days 1, 8, 15 and 22 for five 35-day cycles (Maintenance).
  Interventions: Drug: Bortezomib; Drug: Melphalan; Drug: Prednisone

INTERVENTIONS:
Drug: Bortezomib — Bortezomib bolus intravenous (IV) injection
  Other Names: Velcade
Drug: Dexamethasone — Dexamethasone for oral administration
  Arms: Bortezomib and Dexamethasone (VD); Bortezomib, Thalidomide, and Dexamethasone (VTD)
Drug: Melphalan — Melphalan for oral administration
  Arms: Bortezomib, Melphalan and Prednisone (VMP)
Drug: Prednisone — Prednisone for oral administration
  Arms: Bortezomib, Melphalan and Prednisone (VMP)
Drug: Thalidomide — Thalidomide for oral administration
  Arms: Bortezomib, Thalidomide, and Dexamethasone (VTD)

SUMMARY:
This is a randomized, open label, multicenter clinical trial to compare the efficacy and safety of Velcade (bortezomib) and dexamethasone versus Velcade, thalidomide, and dexamethasone versus Velcade, melphalan, and prednisone in patients with previously untreated multiple myeloma not considered candidates for high-dose chemotherapy and autologous stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years of age or older
* Not a candidate for high-dose chemotherapy and stem cell transplantation (HDT/SCT) due to age, presence of important comorbid condition(s) likely to have a negative impact on tolerability of HDT-SCT, or subject preference.
* A Karnofsky Performance Status score of ≥50%
* Symptomatic multiple myeloma or asymptomatic multiple myeloma with related organ or tissue damage.
* Asymptomatic multiple myeloma-related organ or tissue damage can include presence of an asymptomatic lytic bone lesion or plasmacytoma, the presence of anemia (hemoglobin <10 g/dL), renal function impairment (serum creatinine > upper limit of normal [ULN]) or hypercalcemia (serum calcium >ULN).
* Must have measurable disease requiring systemic therapy. Measurable disease is defined by at least 1 of the following criteria:

  * Quantifiable serum M-protein value (>1 g/dL of immunoglobulin (Ig)G or IgM M-protein, >0.5g/dL of IgA M-protein, >0.5 g/dL of IgD M-protein)
  * Urine light-chain excretion ≥200 mg/24 hours
* Voluntary written informed consent must be given before performance of any study related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the participant at any time without prejudice to future medical care.

Exclusion Criteria:

* Diagnosis of smoldering multiple myeloma or monoclonal gammopathy of undetermined significance (MGUS). Smoldering multiple myeloma is defined as asymptomatic multiple myeloma with absence of lytic bone lesions. MGUS is defined by presence of serum monoclonal protein <3 g/dL; absence of lytic bone lesions, anemia, hypercalcemia, and renal insufficiency related to the monoclonal protein; and (if determined) proportion of plasma cells in the bone marrow of 10% or less.
* Diagnosis of Waldenström's disease or other conditions in which immunoglobulin M (IgM) M-protein is present in the absence of a clonal plasma cell infiltration or lytic bone lesions.
* Previously or currently treated with any systemic therapy for multiple myeloma. Prior treatment of hypercalcemia or spinal cord compression with corticosteroids or radiation therapy, respectively, does not disqualify the subject (the dose of corticosteroids should not exceed the equivalent of 160 mg of dexamethasone in 2-week period).
* Radiation therapy within 2 weeks before randomization. Enrollment of patients who require concurrent radiotherapy (which must be localized in its field size) should be deferred until the radiotherapy is completed and 2 weeks have elapsed since the last date of therapy.
* Major surgery within 30 days before randomization (Kyphoplasty is not considered major surgery)
* History of allergy to any of the study medications, their analogues, or excipients in the various formulations
* ≥Grade 2 peripheral neuropathy on clinical examination within 21 days before enrollment.
* Any of the following clinical laboratory values within 21 days prior to enrollment:

  * Absolute neutrophil count (ANC) <1000 cells/mm^3
  * Platelets <100,000 × 10^9/L, or <70 × 10^9/L if thrombocytopenia is considered by the investigator to be due to myeloma infiltration of bone marrow
  * Aspartate aminotransferase [serum glutamic oxaloacetic transaminase] (AST [SGOT]) or alanine aminotransferase [serum glutamic-pyruvic transaminase] (ALT [SGPT]) >2× the upper limit of normal (ULN)
  * Serum creatinine >2 mg/dL (>176.8 µmol/L); if the rise in creatinine is related to myeloma and there has been demonstrated a response to hydration, the subject may be enrolled.
* Myocardial infarction within 6 months prior to enrollment or New York Hospital Association Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or significant conduction system abnormalities in the opinion of the investigator. Prior to study entry, any abnormality on electrocardiogram at screening must be determined and documented by the investigator as not medically relevant.
* Any condition, including laboratory abnormalities, that in the opinion of the Investigator places the patient at unacceptable risk if he/she were to participate in the study. This includes but is not limited to serious medical conditions or psychiatric illness likely to interfere with participation in this clinical study.
* Prior malignancy except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, in situ breast cancer, in situ prostate cancer, or other cancer for which the patient has been disease-free for at least 3 years.
* Female who is pregnant or breastfeeding. Female participants of childbearing potential must have a negative pregnancy test with a sensitivity of at least 50 mIU/mL during Screening.
* Use of any investigational drugs within 30 days before randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 502 (Actual)
Dates: Start 2007-06; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (234):
- United States (233):
  - Birmingham Hematology Oncology Assciates, LLC, Birmingham, Alabama
  - Desert Oasis Cancer Center, Casa Grande, Arizona
  - Northern Arizona Hematology & Oncology Associates - AOA, Sedona, Arizona
  - Arizona Oncology Associates, Tucson, Arizona
  - Heritage Physician Group Oncology, Hot Springs, Arkansas
  - Hematology Oncology Services of Arkansas, Little Rock, Arkansas
  - Pacific Cancer Medical Centre, Anaheim, California
  - Tower Cancer Research Foundation, Beverly Hills, California
  - Compassionate Cancer Care Medical Group, Corona, California
  - Compassionate Cancer Care Medical Group, Inc., Fountain Valley, California
  - Robert A. Moss, MD, FACP, Inc., Fountain Valley, California
  - Cancer Care Associates, Fresno, California
  - Glendale Memorial Hospital & Health Center, Glendale, California
  - California Cancer Care, Greenbrae, California
  - Beaver Medical Group, Highland, California
  - Edward A. Wagner, MD, Laguna Beach, California
  - Clinical Trials and Research Associates, Inc., Montebello, California
  - Medical Oncology Care Associates, Orange, California
  - Ventura County Hematology Oncology Specialists, Oxnard, California
  - Southwest Cancer Care, Poway, California
  - Desert Cancer Care, Incorporated, Rancho Mirage, California
  - Compassionate Cancer Care Medical Group, Inc., Riverside, California
  - Sutter Cancer Center, Sacramento, California
  - Cancer Research & Prevention Center, Soquel, California
  - Stockton Hematology/Oncology, Stockton, California
  - Trivalley Oncology Hematology, Westlake Village, California
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Cancer Center of Central Connecticut, Southington, Connecticut
  - Christiana Care Health Services, Newark, Delaware
  - The Center for Hematology-Oncology, Boca Raton, Florida
  - Pasco Hernando Oncology, Brooksville, Florida
  - Northwest Oncology & Hematology Associates, Coral Springs, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - Horizon Institute for Clinical Research, Hollywood, Florida
  - Baptist Cancer Institute, Jacksonville, Florida
  - University of Florida- Jacksonville, Jacksonville, Florida
  - Cancer Care of North Florida, Lake City, Florida
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - Cancer & Blood Disease Center, Lecanto, Florida
  - Pasco Hernando Oncology, New Port Richey, Florida
  - Florida Cancer Institute, New Port Richey, Florida
  - Innovative Medical Research of South Florida Inc., North Miami Beach, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Cancer Centers of Florida, P.A., Ocoee, Florida
  - MD Anderson Cancer Center Orlando, Orlando, Florida
  - Hematology Oncology Associates of the Treasure Coast, PA, Port Saint Lucie, Florida
  - Gulfcoast Oncology Associates, St. Petersburg, Florida
  - S. Florida Oncology/ Hematology, West Palm Beach, Florida
  - Medical Oncology Associates of Augusta, Augusta, Georgia
  - Central Georgia Cancer Care, Macon, Georgia
  - Northwest Georgia Oncology Centers, P.C., Marietta, Georgia
  - Summit Cancer Care, Savannah, Georgia
  - St. Lukes Mountain States Tumor Institute, Boise, Idaho
  - Snake River Oncology of Eastern Idaho, PLLC., Idaho Falls, Idaho
  - Cancer Care & Hematology Specialists of Chicagoland, Arlington Heights, Illinois
  - Hematology Oncology Associates of Illinois, Chicago, Illinois
  - John H. Stroger, Jr. Hospital of Cook County, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Oncology Hematology Associates of North Illinois Ltd., Gurnee, Illinois
  - Midwest Center for Hematology / Oncology, Joliet, Illinois
  - Joliet Oncology-Hematology Associates, Ltd., Joliet, Illinois
  - Hematology Oncology Consultants, Inc., Naperville, Illinois
  - Cancer Care and Hematology Specialists of Chicagoland, Niles, Illinois
  - Mid-Illinois Hem & Onc, Normal, Illinois
  - Quincy Medical Group, Quincy, Illinois
  - Deaconess Clinic Incorporated, Evansville, Indiana
  - Central Indiana Cancer Centers, Indianapolis, Indiana
  - Investigative Clinical Research of Indiana, LLC, Indianapolis, Indiana
  - Clarian Arnett Cancer Center, Lafayette, Indiana
  - Medical Consultants, PC, Muncie, Indiana
  - Cancer Care Center, New Albany, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Hope Center, Terre Haute, Indiana
  - McFarland Clinic, P.C., Ames, Iowa
  - Heartland Hematology-Oncology Associates, Inc., Council Bluffs, Iowa
  - Siouxland Hematology/Oncology Assoc., LLP, Sioux City, Iowa
  - Kansas City Cancer Centers - Southwest, Overland Park, Kansas
  - Cancer Center of Kansas, Wichita, Kansas
  - Commonwealth Cancer Center, Danville, Kentucky
  - Kentucky Cancer Clinic, Hazard, Kentucky
  - Western Kentucky Hematology and Oncology Group, Paducah, Kentucky
  - Christus St. Francis Cabrini Cancer Center, Alexandria, Louisiana
  - Hematology-Oncology Clinic, Baton Rouge, Louisiana
  - Annapolis Oncology Center, Annapolis, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - St. Agnes Health Care, Baltimore, Maryland
  - Auerbach Hematology Oncology Associates, Baltimore, Maryland
  - Maryland Hematology Oncology Association, Baltimore, Maryland
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Oncology-Hematology Associates, P.A., Clinton, Maryland
  - Maryland Oncology Hematology, PA, Columbia, Maryland
  - Carroll County Cancer Center, Westminster, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Fallon Clinic at Worcester Medical Center, Worcester, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Cancer & Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - Kalamazoo Hematology and Oncology, Kalamazoo, Michigan
  - Hematology Oncology Associates of Ohio & Michigan, PC, Lambertville, Michigan
  - Breslin Cancer Center / Great Lakes Cancer Institute, Lansing, Michigan
  - Oncology Care Associates, P.L.L.C., Saint Joseph, Michigan
  - Providence Cancer Center, Southfield, Michigan
  - Osteopathic Medical Hematology & Oncology, Woodhaven, Michigan
  - St. Luke's Hospital, Duluth, Minnesota
  - Metro MN CCOP, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center, Robbinsdale, Minnesota
  - St. Louis Cancer Center, Chesterfield, Missouri
  - Capital Region Medical Center/Cancer Center, Jefferson City, Missouri
  - Heartland Hematology-Oncology Associates, Inc., Kansas City, Missouri
  - Kansas City Veterans Administration Medical Center, Kansas City, Missouri
  - St. Joseph Oncology, Saint Joseph, Missouri
  - Great Falls Clinic, LLP, Great Falls, Montana
  - Great Plains Regional Medical Center, North Platte, Nebraska
  - Creighton Cancer Center, Omaha, Nebraska
  - Las Vegas Cancer Center, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Veterans Affairs New Jersey Healthcare System, East Orange, New Jersey
  - Drs. Forte, Schleider, Attas and Condemi, PA, Englewood, New Jersey
  - St. Barnabas Medical Center, Livingston, New Jersey
  - Newark Beth Israel Hospital, Newark, New Jersey
  - Somerset Hematology Oncology Associates, Somerville, New Jersey
  - Sparta Cancer Center, Sparta, New Jersey
  - New Mexico Cancer Care Associates, Santa Fe, New Mexico
  - Stratton VA Medical Center IRB, Albany, New York
  - Buffalo Institute for Medical Research, Inc., Buffalo, New York
  - Erie County Medical Center, Buffalo, New York
  - Goshen Medical Associates, Goshen, New York
  - Huntington Medical Group, Huntington Station, New York
  - North Shore-Long Island Jewish Health System, Lake Success, New York
  - Arena Oncology Associates, New Hyde Park, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital-Cornell Campus, New York, New York
  - Interlakes Foundation, Inc., Rochester, New York
  - Richmond University Medical Center, Staten Island, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Eastchester Center for Cancer Care, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Cancer Care of WNC, Asheville, North Carolina
  - Alamance Regional Medical Center, Burlington, North Carolina
  - Blood and Cancer Clinic, Fayetteville, North Carolina
  - Gaston Hematology & Oncology, Gastonia, North Carolina
  - Carolina Oncology Specialist, PA, Hickory, North Carolina
  - Emerywood Hematology/Oncology, High Point, North Carolina
  - Raleigh Hematology Oncology / Associates, P.C., Raleigh, North Carolina
  - Hanover Medical Specialists, P.A., Wilmington, North Carolina
  - St. Alexius Clinical Research Services, Bismarck, North Dakota
  - Gabrail Cancer Center, Canton, Ohio
  - Oncology Hematology Care, Inc., Cincinnati, Ohio
  - Oncology Partners Network, Cincinnati, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Hematology Oncology Consultants Inc., Columbus, Ohio
  - Dayton Clinical Oncology Program, Dayton, Ohio
  - Dayton Oncology & Hematology, Kettering, Ohio
  - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - Trilogy Cancer Center, Wooster, Ohio
  - Cancer Care Associates, Oklahoma City, Oklahoma
  - Oklahoma Oncology and Hematology, Tulsa, Oklahoma
  - Willamette Valley Cancer Center, Eugene, Oregon
  - Onc-Hem of Lehigh Valley, PC, Bethlehem, Pennsylvania
  - Hematology & Oncology Associates of NEPA, Dunmore, Pennsylvania
  - Medical Oncology Associates, Kingston, Pennsylvania
  - Regional Hematology Oncology Associates, Langhorne, Pennsylvania
  - Greater Philadelphia Cancer and Hematology Specialists, PC, Philadelphia, Pennsylvania
  - UPMC Cancer Pavillioin, Pittsburgh, Pennsylvania
  - Guthrie Research Institute, Sayre, Pennsylvania
  - Scranton Hematology Oncology, Scranton, Pennsylvania
  - Roger Williams Medical Center, Providence, Rhode Island
  - MUSC Hollings Cancer Center, Charleston, South Carolina
  - Cancer Center of the Carolinas, Greenville, South Carolina
  - Low Country Hematology & Oncology, Mt. Pleasant, South Carolina
  - Santee Hematology/Oncology, Sumter, South Carolina
  - Avera Research Institute, Sioux Falls, South Dakota
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - The Family Cancer Center, PLLC, Collierville, Tennessee
  - The Cancer Center of Cookeville Regional Medical Center, Cookeville, Tennessee
  - The Jones Clinic, Germantown, Tennessee
  - East Tennessee Oncology/Hematology, Knoxville, Tennessee
  - University of Tennesee Medical Center, Knoxville, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Texas Cancer Center, Abilene, Texas
  - Texas Oncology, P.A., Arlington, Texas
  - Southwest Regional Cancer Center, Austin, Texas
  - Texas Oncology, PA, Austin, Texas
  - Texas Oncology, PA, Beaumont, Texas
  - Texas Oncology, P.A., Bedford, Texas
  - Coastal Bend Cancer Center, Corpus Christi, Texas
  - South Texas Institute of Cancer and Blood Disorders, Corpus Christi, Texas
  - Texas Oncology, Dallas, Texas
  - Dallas Oncology Consultants, Dallas, Texas
  - Texas Oncology, PA / Methodist Charlton Cancer Center, Dallas, Texas
  - Texas Oncology PA, Dallas, Texas
  - Texas Cancer Center, Denton, Texas
  - El Paso Cancer Treatment Center, El Paso, Texas
  - Texas Cancer Center, Fort Worth, Texas
  - Texas Oncology, PA, Garland, Texas
  - Lee C. Drinkard, MD, Grapevine, Texas
  - Houston Cancer Institute, Houston, Texas
  - Medicus Alliance Clinical Research Organization, LLC, Houston, Texas
  - Lake Vista Cancer Center, Lewisville, Texas
  - Longview Cancer Center, Longview, Texas
  - Texas Cancer Center of Mesquite, Mesquite, Texas
  - Texas Oncology, P.A., Midland, Texas
  - Texas Oncology - Odessa, Odessa, Texas
  - Paris Regional Cancer Center, Paris, Texas
  - Cancer Care Network of South Texas, San Antonio, Texas
  - Cancer Care Center of South Texas, San Antonio, Texas
  - CTRC Institute for Drug Development, San Antonio, Texas
  - Texas Cancer Center - Sherman, Sherman, Texas
  - Blood and Cancer Center of East Texas, Tyler, Texas
  - Tyler Hematology/Oncology, PA, Tyler, Texas
  - Texas Oncology, PA, Tyler, Texas
  - Texas Oncology, Waco, Texas
  - Northern Utah Associates, Ogden, Utah
  - Utah Cancer Specialists, Salt Lake City, Utah
  - The University of Vermont, Burlington, Vermont
  - White River Junction VAMC, White River Junction, Vermont
  - Cancer Specialists of Tidewater, Chesapeake, Virginia
  - Fairfax/Northern Virginia Hematology/Oncology, Fairfax, Virginia
  - Lynchburg Hematology Oncology Clinic, Inc., Lynchburg, Virginia
  - Peninsula Cancer Institute Riverside Cancer Center, Newport News, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Inc., Salem, Virginia
  - Masoom Kandahari, MD, PC, Woodbridge, Virginia
  - Puget Sound Cancer Center - Edmonds, Edmonds, Washington
  - Providence Everett Medical Center, Everett, Washington
  - Puget Sound Cancer Center, Inc, Seattle, Washington
  - Cancer Care Northwest, US Oncology, Spokane, Washington
  - Northwest Medical Specialties, PLLC, Tacoma, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Yakima Valley Memorial Hospital / North Star Lodge, Yakima, Washington
  - Gundersen Clinic, Ltd., La Crosse, Wisconsin
  - Alyce & Elmore Kraemer Cancer Center, West Bend, Wisconsin
- Hospital Auxillo Mutuo, Auxilio Mutuo Cancer Center, San Juan, Puerto Rico

REFERENCES:
- [Derived] Niesvizky R, Flinn IW, Rifkin R, Gabrail N, Charu V, Clowney B, Essell J, Gaffar Y, Warr T, Neuwirth R, Zhu Y, Elliott J, Esseltine DL, Niculescu L, Reeves J. Community-Based Phase IIIB Trial of Three UPFRONT Bortezomib-Based Myeloma Regimens. J Clin Oncol. 2015 Nov 20;33(33):3921-9. doi: 10.1200/JCO.2014.58.7618. Epub 2015 Jun 8. PMID 26056177

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 158 investigative sites in the United States from 26 June 2007 to 28 March 2013
Pre-assignment Details: Participants with previously untreated multiple myeloma were randomized in a 1:1:1 ratio to one of three treatment groups: VD: Velcade (bortezomib) and dexamethasone; VTD: Velcade, thalidomide, and dexamethasone; VMP: Velcade, melphalan, and prednisone.
Groups:
- Bortezomib and Dexamethasone: Participants received bortezomib (Velcade) 1.3 mg/m^2 administered as a bolus intravenous (IV) injection on Days 1, 4, 8, and 11, and dexamethasone 20 mg orally on Days 1, 2, 4, 5, 8, 9, 11 and 12 for eight 21-day treatment cycles (Induction). Participants then received bortezomib 1.6 mg/^2 IV on Days 1, 8, 15 and 22 for five 35-day cycles (Maintenance).
- Bortezomib, Thalidomide, and Dexamethasone: Participants received bortezomib 1.3 mg/m^2 administered as a bolus IV injection on Days 1, 4, 8, and 11, and dexamethasone 20 mg orally on Days 1, 2, 4, 5, 8, 9, 11 and 12, and thalidomide 100 mg orally on Days 1-21 for eight 21-day treatment cycles (Induction). Participants then received bortezomib 1.6 mg/^2 IV on Days 1, 8, 15 and 22 for five 35-day cycles (Maintenance).
- Bortezomib, Melphalan and Prednisone: Participants received bortezomib 1.3 mg/m^2 administered as a bolus IV injection on Days 1, 4, 8, and 11, and melphalan 9 mg/m^2 orally on Days 1-4 every other cycle and prednisone 60 mg/m^2 orally on Days 1-4 every other cycle for eight 21-day treatment cycles (Induction). Participants then received bortezomib 1.6 mg/^2 IV on Days 1, 8, 15 and 22 for five 35-day cycles (Maintenance).
Period: Overall Study
Arm/Group | Bortezomib and Dexamethasone | Bortezomib, Thalidomide, and Dexamethasone | Bortezomib, Melphalan and Prednisone
Started | 168 | 167 | 167
Treated (Safety Population) | 165 | 158 | 163
Completed 8 Treatment Cycles | 82 | 60 | 69
Completed | 50 (Completed is defined as having completed 13 treatment cycles.) | 42 (Completed is defined as having completed 13 treatment cycles.) | 53 (Completed is defined as having completed 13 treatment cycles.)
Not Completed | 118 | 125 | 114
Not completed — Adverse Event | 58 | 67 | 65
Not completed — Protocol Violation | 1 | 2 | 0
Not completed — Lack ofEfficacy / Physician Decision | 7 | 7 | 8
Not completed — Progressive Disease | 20 | 10 | 13
Not completed — Patient declined further treatment | 18 | 14 | 11
Not completed — Other | 11 | 16 | 13
Not completed — Did not Receive Study Treatment | 3 | 9 | 4

BASELINE CHARACTERISTICS:
Population: Intention to treat population, defined as all participants randomized
Groups:
- Total: Total of all reporting groups
Arm/Group | Bortezomib and Dexamethasone | Bortezomib, Thalidomide, and Dexamethasone | Bortezomib, Melphalan and Prednisone | Total
Number analyzed (Participants) | 168 | 167 | 167 | 502
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.6 (9.35) | 71.3 (8.73) | 71.3 (8.67) | 71.7 (8.92)
Age, Customized [Number; unit: participants]
  ≥ 65 years | 140 | 135 | 139 | 414
  ≥ 75 years | 84 | 64 | 62 | 210
  ≥ 80 years | 40 | 27 | 23 | 90
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 97 | 77 | 241
  Male | 101 | 70 | 90 | 261
Race/Ethnicity, Customized [Number; unit: participants]
  White | 131 | 124 | 118 | 373
  Black | 23 | 31 | 29 | 83
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 2 | 2
  Asian | 2 | 1 | 0 | 3
  American Indian or Alaskan Native | 0 | 1 | 2 | 3
  Other | 10 | 10 | 15 | 35
  Not Reported | 2 | 0 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 168 | 167 | 167 | 502

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from randomization to disease progression or death, whichever occurs first. Participants who did not progress and were still alive at the cut-off date were censored at the date of last contact. Response was assessed by the Investigator using the International Myeloma Working Group (IMWG) uniform response criteria.
  Progressive disease requires 1 of the following:
  * Increase of ≥ 25% from nadir in:
    * Serum M-component (absolute increase ≥ 0.5 g/dl)
    * Urine M-component (absolute increase ≥ 200 mg/24 hours)
    * In patients without measurable serum and urine M-protein levels the difference between involved and uninvolved free light chain (FLC) levels (absolute increase > 100 mg/dl)
    * Bone marrow plasma cell percentage (absolute % ≥ 10%)
  * Development of new or increase in the size of existing bone lesions or soft tissue plasmacytomas.
  * Development of hypercalcemia (corrected serum calcium > 11.5 mg/dl) attributed solely to plasma cell proliferative disease
Time Frame: From randomization until disease progression. Median follow-up time was 43 months.
Population: Intent-to-treat (all randomized participants)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bortezomib and Dexamethasone | Bortezomib, Thalidomide, and Dexamethasone | Bortezomib, Melphalan and Prednisone
Number analyzed (Participants) | 168 | 167 | 167
months | 14.7 [12.0 to 18.6] | 15.4 [12.6 to 24.2] | 17.3 [14.8 to 20.3]
Statistical Analysis 1: Comparison: Bortezomib and Dexamethasone vs Bortezomib, Thalidomide, and Dexamethasone vs Bortezomib, Melphalan and Prednisone; Test type: Superiority or Other; p = 0.458, Wald test — The global difference among arms was based on the Wald test

2. Secondary Outcome: Percentage of Participants With an Overall Response
Description: Overall response defined as a best overall response of complete response (CR), very good partial response (VGPR) or partial response (PR), assessed by the Investigator using the IMWG uniform response criteria.
  CR: Negative immunofixation on the serum and urine, disappearance of any soft tissue plasmacytomas, and <5% plasma cells in bone marrow.
  VGPR: Serum and urine M-protein detectable by immunofixation but not on electrophoresis or ≥ 90% reduction in serum M-protein plus urine M-protein level <100 mg per 24 hours (h).
  PR requires 1 of the following:
  * ≥50% reduction of serum M-protein and 24-h urinary M-protein by ≥ 90% or to <200 mg/24 h, or
  * If M-protein not measurable, a ≥50% decrease in the difference between involved and uninvolved FLC levels, or
  * If FLC not measurable, a ≥ 50% reduction in plasma cells, provided baseline bone marrow plasma cell percentage was ≥30%.
  If present at baseline, a ≥50% reduction in the size of soft tissue plasmacytomas is also required.
Time Frame: Response assessed every other cycle for up to 13 cycles (49 weeks).
Population: Response-Evaluable population, defined as all participants who received at least 1 dose of any study drug, have measurable disease at baseline, and have at least one post-baseline M-protein measurement.
Measure: Number; unit: percentage of participants
Arm/Group | Bortezomib and Dexamethasone | Bortezomib, Thalidomide, and Dexamethasone | Bortezomib, Melphalan and Prednisone
Number analyzed (Participants) | 147 | 133 | 145
percentage of participants | 73 | 80 | 70

3. Secondary Outcome: Percentage of Participants With a Complete Response
Description: Participants with a best overall response of complete response, defined as negative immunofixation on the serum and urine, disappearance of any soft tissue plasmacytomas, and <5% plasma cells in bone marrow. Response was assessed by the Investigator using the IMWG uniform response criteria.
Time Frame: Response assessed every other cycle, for up to 13 cycles (49 weeks).
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Bortezomib and Dexamethasone | Bortezomib, Thalidomide, and Dexamethasone | Bortezomib, Melphalan and Prednisone
Number analyzed (Participants) | 147 | 133 | 145
percentage of participants | 3 | 4 | 4

4. Secondary Outcome: Percentage of Participants With a Complete Response or a Very Good Partial Response
Description: Complete response is defined by negative immunofixation on the serum and urine, disappearance of any soft tissue plasmacytomas, and <5% plasma cells in bone marrow.
  Very good partial response is defined by serum and urine M-protein detectable by immunofixation but not on electrophoresis or 90% or greater reduction in serum M-protein plus urine M-protein level <100 mg per 24 hours.
  Response was assessed by the Investigator using the IMWG uniform response criteria.
Time Frame: Response assessed every other cycle for up to 13 cycles (49 weeks).
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Bortezomib and Dexamethasone | Bortezomib, Thalidomide, and Dexamethasone | Bortezomib, Melphalan and Prednisone
Number analyzed (Participants) | 147 | 133 | 145
percentage of participants | 37 | 51 | 41

5. Secondary Outcome: Duration of Response
Description: Duration of response is defined in participants with an overall response as the time between first documentation of response and disease progression. Responders without disease progression were censored at the last clinical assessment of response.
Time Frame: From first documented response until disease progression. Median follow-up time was 43 months.
Population: Participants with an overall response
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bortezomib and Dexamethasone | Bortezomib, Thalidomide, and Dexamethasone | Bortezomib, Melphalan and Prednisone
Number analyzed (Participants) | 107 | 106 | 101
months | 18.3 [14.3 to 24.2] | 22.4 [12.7 to 29.1] | 19.8 [16.4 to 23.3]

6. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time between randomization and death. Participants still alive at the cutoff date or lost to follow-up were censored at the date of last contact.
Time Frame: From randomization until death. Median follow-up time was 43 months.
Population: Intent to treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bortezomib and Dexamethasone | Bortezomib, Thalidomide, and Dexamethasone | Bortezomib, Melphalan and Prednisone
Number analyzed (Participants) | 168 | 167 | 167
months | 49.8 [35.7 to NA] — Upper limit was not estimable due to low number of events | 51.5 [38.5 to NA] — Upper limit was not estimable due to low number of events | 53.1 [41.1 to NA] — Upper limit was not estimable due to low number of events

7. Secondary Outcome: Time to Alternative Therapy
Description: Time to alternative therapy is defined as the time between randomization and alternative therapy. Participants who did not receive alternative therapy were censored at the time of last contact.
Time Frame: From randomization until alternative therapy. Median follow-up time was 43 months.
Population: Intent to Treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bortezomib and Dexamethasone | Bortezomib, Thalidomide, and Dexamethasone | Bortezomib, Melphalan and Prednisone
Number analyzed (Participants) | 168 | 167 | 167
months | 19.7 [16.0 to 27.8] | 24.5 [16.6 to 27.6] | 19.0 [15.2 to 23.1]

8. Secondary Outcome: Change From Baseline in EORTC QLQ-C30 - Global Health Status
Description: The European Organisation for Research and Treatment of Cancer (EORTC) Core Quality of Life (QOL) questionnaire (EORTC QLQ-C30) is a 30-question tool used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact).
  The EORTC QLQ-C30 Global Health Status/QOL Scale is scored between 0 and 100, where higher scores indicate better Global Health Status/QOL. Negative changes from baseline indicate deterioration in QOL or functioning and positive changes indicate improvement.
Time Frame: Baseline and Day 1 of Cycles 3, 5, 7, 9, 11 and 13
Population: Intent-to-treat population with available data at each time point (indicated by "n").
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bortezomib and Dexamethasone | Bortezomib, Thalidomide, and Dexamethasone | Bortezomib, Melphalan and Prednisone
Number analyzed (Participants) | 168 | 167 | 167
units on a scale
  Cycle 3, Day 1 (n=129, 115, 125) | 1.3 (25.40) | -4.4 (27.04) | 2.0 (30.82)
  Cycle 5, Day 1 (n=114, 98, 107) | -4.9 (30.36) | -6.1 (27.47) | -0.4 (29.24)
  Cycle 7, Day 1 (n=89, 79, 84) | -3.3 (32.58) | -8.6 (31.86) | -4.7 (28.61)
  Cycle 9, Day 1 (n=87, 66, 67) | -4.2 (33.55) | -8.1 (28.16) | -1.0 (28.55)
  Cycle 11, Day 1 (n=71, 61, 65) | -11.6 (33.67) | -7.9 (29.54) | 2.8 (31.72)
  Cycle 13, Day 1 (n=67, 52, 61) | -10.2 (36.00) | -8.5 (32.87) | 1.0 (35.16)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the first dose of study drug through 30 days after the last dose of study drug. Treatment was administered for up to 49 weeks.
Description: Per protocol, all grades of peripheral neuropathy and skeletal events, Grade 3/4 AEs, and all SAEs were recorded. There may be grade 1 or 2 events that were not required to be collected.
Arm/Group | Bortezomib and Dexamethasone | Bortezomib, Thalidomide, and Dexamethasone | Bortezomib, Melphalan and Prednisone
Serious Adverse Events (participants affected / at risk) | 88/165 | 92/158 | 83/163
Other Adverse Events (participants affected / at risk) | 57/165 | 68/158 | 68/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bortezomib and Dexamethasone (N=165) | Bortezomib, Thalidomide, and Dexamethasone (N=158) | Bortezomib, Melphalan and Prednisone (N=163)
Pneumonia (Infections and infestations) | 18 | 12 | 10
Lobar pneumonia (Infections and infestations) | 1 | 2 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 3 | 1 | 2
Bacteraemia (Infections and infestations) | 1 | 1 | 2
Septic shock (Infections and infestations) | 0 | 2 | 0
Bacterial sepsis (Infections and infestations) | 0 | 1 | 0
Device related sepsis (Infections and infestations) | 1 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 2 | 4
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 2
Diverticulitis (Infections and infestations) | 0 | 1 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 3 | 1 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 1 | 0
Peritonitis bacterial (Infections and infestations) | 0 | 1 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 2
Herpes zoster disseminated (Infections and infestations) | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 1 | 1
Staphylococcal abscess (Infections and infestations) | 0 | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0 | 0
Bursitis infective (Infections and infestations) | 0 | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 1 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 0 | 1
Device related infection (Infections and infestations) | 1 | 0 | 0
Pneumonia pneumococcal (Infections and infestations) | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 12 | 5 | 8
Vomiting (Gastrointestinal disorders) | 3 | 5 | 6
Nausea (Gastrointestinal disorders) | 2 | 4 | 4
Constipation (Gastrointestinal disorders) | 6 | 3 | 3
Abdominal pain (Gastrointestinal disorders) | 4 | 3 | 4
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 4 | 1
Ileus (Gastrointestinal disorders) | 1 | 1 | 3
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0
Large intestinal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Duodenal perforation (Infections and infestations) | 0 | 0 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 1 | 0
Gastric perforation (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 8 | 6 | 9
Hypovolaemia (Metabolism and nutrition disorders) | 2 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 1 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 3 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 2 | 5 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 3 | 0
Peripheral motor neuropathy (Nervous system disorders) | 2 | 1 | 0
Neuralgic amyotrophy (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 5 | 5 | 5
Lethargy (Nervous system disorders) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0
Spinal haematoma (Nervous system disorders) | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 2 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 1
Dizziness postural (Nervous system disorders) | 1 | 0 | 0
Dementia (Nervous system disorders) | 0 | 1 | 0
Dementia with Lewy bodies (Nervous system disorders) | 0 | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 1 | 0
VIth nerve paralysis (Nervous system disorders) | 0 | 0 | 1
Sciatica (Nervous system disorders) | 1 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 1
Quadriplegia (Nervous system disorders) | 0 | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 1 | 0
Asthenia (General disorders) | 6 | 3 | 3
Fatigue (General disorders) | 1 | 4 | 2
Pyrexia (General disorders) | 7 | 2 | 2
Pain (General disorders) | 0 | 1 | 2
Chest pain (General disorders) | 1 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 2 | 0
Oedema peripheral (General disorders) | 1 | 2 | 1
Generalised oedema (General disorders) | 0 | 1 | 0
Death (General disorders) | 2 | 1 | 1
Multi-organ failure (General disorders) | 1 | 0 | 1
Chills (General disorders) | 0 | 0 | 1
Nodule (General disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 7 | 7 | 1
Atrial flutter (Cardiac disorders) | 3 | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 7 | 8 | 1
Angina pectoris (Cardiac disorders) | 1 | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 2 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1
Right ventricular failure (Cardiac disorders) | 0 | 1 | 0
Tricuspid valve incompetence (Cardiac disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 3 | 3 | 6
Orthostatic hypotension (Cardiac disorders) | 5 | 1 | 5
Deep vein thrombosis (Vascular disorders) | 7 | 4 | 2
Jugular vein thrombosis (Vascular disorders) | 1 | 0 | 0
Peripheral embolism (Vascular disorders) | 0 | 0 | 1
Shock haemorrhagic (Vascular disorders) | 0 | 0 | 1
Phlebitis (Vascular disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 3 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 3 | 5 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Brain contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Extradural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0
Fractured ischium (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 1 | 0
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 | 0 | 1
Drug dispensing error (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 4 | 6 | 2
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 3
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 2 | 1 | 3
Renal failure acute (Renal and urinary disorders) | 1 | 2 | 2
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 2 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1
Renal tubular necrosis (Renal and urinary disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
International normalised ratio increased (Investigations) | 1 | 1 | 1
Prothrombin time prolonged (Investigations) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0 | 1
Klebsiella test positive (Investigations) | 0 | 0 | 1
Blood culture positive (Investigations) | 0 | 0 | 1
Blood potassium decreased (Investigations) | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0
Troponin I increased (Investigations) | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 1
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0 | 1
Depression (Psychiatric disorders) | 1 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 2 | 0
Panic attack (Psychiatric disorders) | 0 | 1 | 0
Acute psychosis (Psychiatric disorders) | 0 | 1 | 0
Withdrawal syndrome (Psychiatric disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 1 | 0
Hepatitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bortezomib and Dexamethasone (N=165) | Bortezomib, Thalidomide, and Dexamethasone (N=158) | Bortezomib, Melphalan and Prednisone (N=163)
Weight decreased (Investigations) | 4 | 2 | 6
Platelet count decreased (Investigations) | 3 | 1 | 7
Blood sodium decreased (Investigations) | 3 | 3 | 3
Blood uric acid increased (Investigations) | 2 | 3 | 3
Neutrophil count decreased (Investigations) | 0 | 0 | 6
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 3
Blood urea increased (Investigations) | 1 | 1 | 1
Protein total increased (Investigations) | 1 | 1 | 1
Weight increased (Investigations) | 0 | 3 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 1
Troponin T increased (Investigations) | 1 | 0 | 1
Blood calcium increased (Investigations) | 0 | 1 | 0
Blood chloride decreased (Investigations) | 0 | 0 | 1
Blood creatinine decreased (Investigations) | 0 | 0 | 1
Blood glucose increased (Investigations) | 0 | 1 | 0
Blood immunoglobulin G increased (Investigations) | 1 | 0 | 0
Blood phosphorus decreased (Investigations) | 0 | 1 | 0
Blood potassium increased (Investigations) | 0 | 1 | 0
Breath sounds abnormal (Investigations) | 0 | 1 | 0
Carbon monoxide diffusing capacity decreased (Investigations) | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 1
Lymphocyte count increased (Investigations) | 1 | 0 | 0
Red blood cell count decreased (Investigations) | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 2 | 4 | 2
Post herpetic neuralgia (Nervous system disorders) | 2 | 2 | 1
Tremor (Nervous system disorders) | 2 | 2 | 1
Balance disorder (Nervous system disorders) | 2 | 2 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 3
Headache (Nervous system disorders) | 1 | 1 | 1
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 | 1 | 2
Somnolence (Nervous system disorders) | 1 | 2 | 0
Ageusia (Nervous system disorders) | 1 | 0 | 1
Cranial nerve disorder (Nervous system disorders) | 0 | 2 | 0
Dysarthria (Nervous system disorders) | 0 | 2 | 0
Memory impairment (Nervous system disorders) | 1 | 1 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 1 | 0
Hypogeusia (Nervous system disorders) | 0 | 1 | 0
Polyneuropathy (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 5 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 4
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Heat rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 9 | 6 | 6
Anxiety (Psychiatric disorders) | 1 | 1 | 1
Mood altered (Psychiatric disorders) | 2 | 1 | 0
Disorientation (Psychiatric disorders) | 1 | 1 | 0
Mood swings (Psychiatric disorders) | 2 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0
Anhedonia (Psychiatric disorders) | 0 | 1 | 0
Anxiety disorder due to a general medical condition (Psychiatric disorders) | 0 | 1 | 0
Delusion (Psychiatric disorders) | 0 | 1 | 0
Depressed mood (Psychiatric disorders) | 1 | 0 | 0
Dysphoria (Psychiatric disorders) | 0 | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 0
Restlessness (Psychiatric disorders) | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 4
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 2
Conjunctivitis bacterial (Infections and infestations) | 0 | 2 | 0
Hordeolum (Infections and infestations) | 0 | 2 | 0
Oral fungal infection (Infections and infestations) | 0 | 1 | 1
Sinusitis (Infections and infestations) | 1 | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 1
Furuncle (Infections and infestations) | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0
Herpes zoster ophthalmic (Infections and infestations) | 0 | 1 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0
Pneumococcal sepsis (Infections and infestations) | 1 | 0 | 0
Skin bacterial infection (Infections and infestations) | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 3 | 8 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 1 | 12
Lymphopenia (Blood and lymphatic system disorders) | 0 | 2 | 4
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Vision blurred (Eye disorders) | 3 | 5 | 1
Conjunctivitis (Eye disorders) | 1 | 2 | 1
Eye swelling (Eye disorders) | 2 | 0 | 0
Visual impairment (Eye disorders) | 0 | 2 | 0
Blepharitis (Eye disorders) | 1 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 1 | 0
Diplopia (Eye disorders) | 0 | 1 | 0
Eye haemorrhage (Eye disorders) | 0 | 0 | 1
Eye pruritus (Eye disorders) | 0 | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 3 | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck mass (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Gait disturbance (General disorders) | 0 | 1 | 2
Catheter site erythema (General disorders) | 0 | 0 | 1
Drug withdrawal syndrome (General disorders) | 0 | 1 | 0
Face oedema (General disorders) | 0 | 1 | 0
Feeling jittery (General disorders) | 0 | 1 | 0
Influenza like illness (General disorders) | 1 | 0 | 0
Irritability (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0
Oedema (General disorders) | 0 | 1 | 0
Soft tissue inflammation (General disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 3 | 2
Hot flush (Vascular disorders) | 1 | 0 | 1
Haematoma (Vascular disorders) | 1 | 0 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1 | 0
Withdrawal hypertension (Vascular disorders) | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 2 | 0 | 3
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 2
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 1
Azotaemia (Renal and urinary disorders) | 0 | 0 | 1
Nocturia (Renal and urinary disorders) | 1 | 0 | 0
Avulsion fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 0 | 1
Restrictive cardiomyopathy (Cardiac disorders) | 0 | 0 | 1
Sick sinus syndrome (Cardiac disorders) | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 2 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0
Cushingoid (Endocrine disorders) | 0 | 1 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi-site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.